CLINICAL TRIAL: NCT04560075
Title: ETUDES Center- Text2Connect - Phase 2
Brief Title: Text 2 Connect- Texting Intervention for Mental Health Treatment Utilization
Acronym: T2C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Kaiser Foundation Research Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tina R Goldstein, Associate Professor of Psychiatry and Psychology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY20060206; P50MH115838-02 (NIH)
Record Dates: First submitted 2020-09-10; First posted 2020-09-23 (Actual); Results first posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Depression; Suicidal Ideation
Keywords: depression; suicidal ideation; treatment; mental health; text message intervention
MeSH Terms: conditions — Depression; Suicidal Ideation; Psychological Well-Being | interventions — Single Person

STUDY DESIGN:
Intervention Model Description: This study will use a parallel study design, where participants are randomized into two intervention groups (T2C and PE) and will receive interventions in parallel.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be masked to the intervention condition at follow-up assessment time points.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text2Connect (Experimental): Participants receiving Text2Connect (T2C) personalized messages will receive a monthly check-in text prompt. Based on their response, the participants then receive either general psychoeducational videos and prompts to continue to monitor mental health or are then prompted to endorse stressors and symptoms they are experiencing to prompt awareness of treatment targets in daily life.
  Interventions: Behavioral: Text2Connect
- Psychoeducational Videos (PE) Only (Active Comparator): Participants will receive a web link to a library of 4 PE videos. These brief 2-minute videos include general information about self-care during college.
  Interventions: Behavioral: Psychoeducational Videos (PE) Only

INTERVENTIONS:
Behavioral: Text2Connect — The T2C intervention aims to increase mental health self-efficacy though psychoeducation, self-monitoring of symptoms and stressors, and cues to action for college-bound youth.
  Arms: Text2Connect
Behavioral: Psychoeducational Videos (PE) Only — Participants in this group will receive psychoeducation through the PE video library.
  Arms: Psychoeducational Videos (PE) Only

SUMMARY:
Text2Connect (T2C) proposes to test a text-based intervention designed to improve engagement with mental health treatment.

DETAILED DESCRIPTION:
To enhance outcomes for transition-age youth with mental health disorders during the vulnerable period that occurs during their first several months of college, the investigators propose an automated TM intervention, "Text to Connect" (T2C), that aims to increase mental health self-efficacy through psychoeducation, self-monitoring of symptoms and stressors, and cues to action for college-bound youth.

Assignment of Interventions:

The study will utilize block randomization whereby 2/3 of participants will be randomly assigned to receive T2C, and 1/3 to receive PE. Blocks will balance the groups on site (CCP versus STAR/CABS). A 2:1 randomization scheme will randomize 50 youth to either receive T2C (n=30) or a link to brief psychoeducational videos about mental health (PE; n=20). All participants will then complete a brief battery of self-report assessments online at baseline and again monthly through month 4. Youth randomized to receive PE will receive a text message with the link to the webpage with the psychoeducational videos. Youth randomized to receive T2C will be onboarded and initiate the TM intervention that sends automated prompts at minimum monthly through month 4.

Hypothesis:

Aim 1. To examine the feasibility of T2C for transition-age youth with psychiatric disorders (n=3 clinics, 50 adolescents). Youth randomized to receive T2C will:

Hypothesis 1a. engage with T2C at high rates (>70% response rate to SMS prompts).

Hypothesis 1b. report high levels of satisfaction (>70% satisfaction) and usability with T2C.

Aim 2. To examine the impact of T2C versus PE on mental health self-efficacy, symptoms and functioning, and treatment engagement. Over 4 months, youth who receive T2C, as compared with youth who receive PE, will report:

Hypothesis 2a (Primary). Greater mental health self-efficacy Hypothesis 2b (Secondary). Lower symptom severity and greater psychosocial functioning Hypothesis 2c (Secondary). Higher rates of follow-through with mental health services

ELIGIBILITY:
Inclusion Criteria:

* Participant engaged in treatment at CC Waterdam, STAR or CABS clinic
* Participants have a current psychiatric diagnosis documented in their electronic medical record and/or be in receipt of mental health services within 3 months per self-/ parent- or clinician- report
* At least 18 years of age
* Recently graduated high school
* Planning to attend college or higher education program within 6 weeks
* Own a text-capable phone
* Be willing and able to provide informed consent

Exclusion Criteria:

* Participants will be excluded if they have conditions that might impair their ability to effectively engage in Text2Connect
* Under the age of 18yo
* Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Goldstein, PhD, Principal Investigator — University of Pittsburgh; Brian Suffoletto, MD, Study Director — University of Pittsburgh Medical Center
Locations (3):
- United States (3):
  - Children's Community Pediatrics (CCP- Waterdam) of Children's Hospital of Pittsburgh UPMC, McMurray, Pennsylvania
  - Child and Adolescent Bipolar Spectrum Services (CABS) Center, Pittsburgh, Pennsylvania
  - STAR Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All requests for study data will follow NIMH's data sharing and data use policies. The final completely de-identified dataset(s) will include demographic and clinical data at baseline, and primary and secondary outcomes for all studies, including those funded by the innovation contests. These analytic datasets may also include derived variables with documentation. Our form datasets will include original case report forms, a detailed codebook of variable names, value labels, and programming formats and all study documentation including the protocol and manual of procedures. For descriptive/raw data, study investigators/study staff will upload to NIMH's National Database for Clinical Trials Related to Mental Health Illness (NDCT) on a semi-annual basis all analyzed data being uploaded prior to primary paper publication.
Time Frame: These data will be released to the NDCT soon after each project's "main outcomes" manuscript is accepted for publication
Access Criteria: In addition to public access to the NDCT, data can also be accessed by contacting ETUDES Center investigators.

REFERENCES:
- [Derived] Suffoletto B, Goldstein T, Gotkiewicz D, Gotkiewicz E, George B, Brent D. Acceptability, Engagement, and Effects of a Mobile Digital Intervention to Support Mental Health for Young Adults Transitioning to College: Pilot Randomized Controlled Trial. JMIR Form Res. 2021 Oct 14;5(10):e32271. doi: 10.2196/32271. PMID 34647893

RESULTS

PARTICIPANT FLOW:
Groups:
- Text2Connect Intervention: Participants receiving Text2Connect (T2C) personalized messages will receive a monthly check-in text prompt. Based on their response, the participants then receive either general psychoeducational videos and prompts to continue to monitor mental health or are then prompted to endorse stressors and symptoms they are experiencing to prompt awareness of treatment targets in daily life.
  Text2Connect: The T2C intervention aims to increase mental health self-efficacy though psychoeducation, self-monitoring of symptoms and stressors, and cues to action for college-bound youth.
- Usual Care-Psychoeducational Videos (PE) Only: Participants will receive a web link to a library of 4 PE videos. These brief 2-minute videos include general information about self-care during college.
  Psychoeducational Videos (PE) Only: Participants in this group will receive psychoeducation through the PE video library.
Period: Overall Study
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Started | 34 | 18
Completed | 34 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only | Total
Number analyzed (Participants) | 34 | 18 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 18 | 52
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 18 | 45
  Male | 7 | 0 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 32 | 17 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 33 | 15 | 48
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Mental health self-efficacy [Mean (Standard Deviation); unit: score on a scale] — Mental health self-efficacy will be assessed via the Mental Health Self-Efficacy Scale (MHSES), as the primary outcome of Text2Connect Phase 2. The MHSES contains 6 items that are scored on a 10-point Likert Scale. Scores range from 6-60 with higher scores indicating greater confidence in participant's mental health self-efficacy.
  score on a scale | 40.3 (10.7) | 37.4 (12.0) | 39.3 (11.1)
General self-efficacy [Mean (Standard Deviation); unit: score on a scale] — Mental health self-efficacy will be assessed via the General Self-Efficacy Scale (GSE), as the primary outcome of Text2Connect Phase 2. The GSE contains 10 items scored on a 4-point Likert Scale, with scores ranging from 10-40. Higher scores indicate greater self-efficacy.
  score on a scale | 29.5 (3.9) | 27.5 (3.3) | 28.8 (3.8)
Symptom Severity [Mean (Standard Deviation); unit: score on a scale] — Symptom severity will be assessed via the CCAPS Mental Health Symptoms. The CCAPS is a 62-item instrument with 8 subscales (depression, general anxiety, social anxiety, academic distress, eating concerns, family distress, hostility, substance abuse) related to psychological symptoms & distress in college students. Scores are on a 5 point likert scale for each subscale: 0 (not at all like me), 1,2,3,4 (Extremely like me). Lower scores indicate greater severity of symptoms. Some items are reverse-scored. To score, average the items scores for each subscale to create the subscale raw score.
  score on a scale
    Depression | 1.43 (0.95) | 1.81 (0.99) | 1.56 (0.97)
    General Anxiety | 1.80 (0.98) | 2.22 (0.95) | 1.94 (0.98)
    Social Anxiety | 2.11 (0.93) | 2.37 (0.93) | 2.20 (0.93)
    Academic Distress | 1.42 (1.02) | 1.90 (0.88) | 1.58 (1.00)
    Eating Concerns | 1.37 (0.89) | 1.51 (1.06) | 1.42 (0.94)
    Family Distress | 1.28 (0.85) | 1.58 (0.81) | 1.39 (0.84)
    Hostility | 1.00 (0.83) | 1.38 (0.61) | 1.13 (0.78)
    Substance Abuse | 0.33 (0.60) | 0.33 (0.72) | 0.33 (0.64)
Mental health service follow-through [Count of Participants; unit: Participants] — Mental health service follow-through will be assessed via the Client Service Receipt Inventory (CSRI). Ratings of 4 questions are Yes or No indicating if participants received the type of service. Scores described below are count of participants indicating "Yes" on the scale.
  Participants
    Any mental health | 19 | 12 | 31
    Inpatient | 2 | 2 | 4
    Outpatient | 13 | 9 | 22
    Primary Care | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Engagement With Intervention: Text Message Check-ins
Description: Participant's engagement with the T2C intervention will be assessed via their response rate to SMS prompts, as the primary outcome of Text2Connect Phase 2. "High" engagement with T2C will be rated as >70% response rate.
  All Intervention participants (n=34) received text-message check-ins with question: "How would you rate your emotional health this past week?" on a likert scale of: 1=excellent; 2=very good; 3=good;4=fair; 5=poor. Participants who did not respond to this message initially were sent a reminder with the same content each week of the intervention.
Time Frame: Over 3 months after baseline
Population: 2 participants lost to follow up at 1 month timepoint after baseline, 1 additional participant lost to follow up 3 month time point with final 31/34 participants completing research visits.
Measure: Median (Full Range); unit: # of text messages sent to participants
Arm/Group | Text2Connect Intervention
Number analyzed (Participants) | 34
# of text messages sent to participants | 5 [3 to 10]

2. Primary Outcome: Engagement With Intervention: Web-based Check Ins
Description: Participant's engagement with the T2C intervention will be assessed via their response rate to prompts, as the primary outcome of Text2Connect Phase 2. "High" engagement with T2C will be rated as >70% response rate.
  Participants received 1 text "How would you rate our emotional health this last week" on a likert scale of: 1 (excellent), 2 Very good, 3 good 4 fair 5 poor. If respondents answered "fair" or "Poor" they were routed to a website with psychoeducational videos and additional questions called a "web-based check in." The questions inquired what type of stressors the participant experienced contributing to the "Fair" or "Poor" ratings, what types of symptoms the participants noticed as a result of the indicated stressor and if participants felt they could manage their stress.
Time Frame: Over 3 months after baseline
Population: 2 participants lost to follow up at 1 month timepoint after baseline, 1 additional participant lost to follow up 3 month time point with final 31/34 participants completing research visits.
  21/34 participants in this arm reported poor mental health on text-messages and therefore were provided with these web-based check ins.
Measure: Count of Units; unit: total number of web-based check-ins
Units Other Than Participants: total number of web-based check-ins
Arm/Group | Text2Connect Intervention
Number analyzed (Participants) | 21
Number analyzed (total number of web-based check-ins) | 55
total number of web-based check-ins | 43

3. Primary Outcome: Engagement With Intervention: Drop Out Rate
Description: Participant's engagement with the T2C intervention will be assessed via their response rate to prompts, as the primary outcome of Text2Connect Phase 2. "High" engagement with T2C will be rated as >70% response rate. Participants are considered "dropped out" if they requested to be removed from the T2C intervention and all texts to be stopped.
Time Frame: Over 3 months after baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Text2Connect Intervention
Number analyzed (Participants) | 34
Participants | 0

4. Primary Outcome: Usability & Satisfaction-PSSUQ
Description: Satisfaction with the technical components of interventions will be assessed through the certain questions from the Post System Satisfaction and Usability Questionnaire (PSSUQ), as the primary outcome of Text2Connect Phase 2. The PSSUQ utilize 16 items w/ response options ranging from 1-7 where 1=strongly disagree and 7=strongly agree. The PSSUQ has sub-scores derived from subsets of the questions which reflect system usefulness, information quality, and interface quality. Scores are added and range from 16-112, with higher score indicating less satisfaction. Questions 1 to 16 result in the Overall score; Questions 1 to 6 result in System Usefulness score; Questions 7 to 12 result in Information Quality score; Questions 13 to 16 result in Interface Quality.
Time Frame: 3 month follow up timepoint
Population: In Intervention Arm: 2 participants lost to follow up at 1 month timepoint after baseline, 1 additional participant lost to follow up 3 month time point with final 31/34 participants completing research visits.
  In Usual Care Arm: 1 participant lost to follow up at 1 month time point, 2 additional participants lost to follow up at 2 month time point and 1 further participant lost at 3 month follow up timepoint. A total of 14/18 completed research visits in usual care arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 31 | 14
score on a scale
  Overall Score | 32.3 (25.3) | 35.4 (25.2)
  System usefulness | 11.4 (9.9) | 12.0 (8.4)
  Quality of information | 13.1 (9.0) | 14.4 (10.3)
  Quality of interface | 7.7 (6.7) | 9.0 (7.3)

5. Primary Outcome: Usability & Satisfaction-CSQ
Description: Satisfaction with the technical components of interventions will be assessed through the certain questions from the Client Satisfaction Questionnaire (CSQ8). 8 items are scored on a likert scale of 1 to 4. Item 1 (reverse scored): scale 1(excellent)-4 (poor); Item 2: 1(definitely not)-4(definitely); item 3(reverse scored): 1(none of needs met)-4(all needs met); item 4: 1(definitely not)-4(definitely); item 5: 1(quite dissatisfied)-4(very satisfied); item 6(reverse scored): 1(made things worse)-4(helped a great deal); item 7 (reverse scored): 1(quite dissatisfied)-4(very satisfied); item 8: 1(definitely not)-4(definitely). Higher scores=higher satisfaction (score sum range is 8-32).
Time Frame: 3 month follow up timepoint
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 31 | 14
score on a scale | 27.4 (4.1) | 25.4 (5.8)

6. Primary Outcome: Mental Health Self-Efficacy
Description: Mental health self-efficacy will be assessed via the Mental Health Self-Efficacy Scale (MHSES), as the primary outcome of Text2Connect Phase 2. The MHSES contains 6 items that are scored on a 10-point Likert Scale. Scores range from 6-60 with higher scores indicating greater confidence in participant's mental health self-efficacy.
Time Frame: 1 month timepoint
Population: In Intervention Arm: 2 participants lost to follow up at 1 month timepoint after baseline
  In Usual Care Arm: 1 participant lost to follow up at 1 month time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 32 | 17
score on a scale | 42.6 (11.2) | 37.9 (11.0)

7. Primary Outcome: Mental Health Self-Efficacy
Description: as for outcome 6
Time Frame: 3 month timepoint
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 31 | 14
score on a scale | 44.0 (11.0) | 39.5 (12.4)

8. Primary Outcome: Mental Health Self-Efficacy
Description: as for outcome 6
Time Frame: 2 month timepoint
Population: In Intervention Arm: 2 participants lost to follow up at 1 month timepoint after baseline
  Usual Care: 2 additional participants lost to follow up at 2 month time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 32 | 15
score on a scale | 42.9 (11.3) | 39.9 (10.7)

9. Primary Outcome: General Self-Efficacy
Description: Mental health self-efficacy will be assessed via the General Self-Efficacy Scale (GSE), as the primary outcome of Text2Connect Phase 2. The GSE contains 10 items scored on a 4-point Likert Scale, with scores ranging from 10-40. Higher scores indicate greater self-efficacy.
Time Frame: 1 month Timepoint
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 32 | 17
score on a scale | 29.7 (4.4) | 28.3 (3.8)

10. Primary Outcome: General Self-Efficacy
Description: as for outcome 9
Time Frame: 2 month Timepoint
Population: In Intervention Arm: 2 participants lost to follow up at 1 month timepoint after baseline
  In Usual Care Arm: 1 participant lost to follow up at 1 month time point, 2 additional participants lost to follow up at 2 month time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 32 | 15
score on a scale | 30.0 (4.2) | 27.6 (4.7)

11. Primary Outcome: General Self-Efficacy
Description: as for outcome 9
Time Frame: 3 month Timepoint
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 31 | 14
score on a scale | 31.3 (5.2) | 27.2 (4.1)

12. Secondary Outcome: Psychosocial Functioning
Description: Psychosocial functioning will be assessed via the College Adjustment Questionnaire (CAQ) The CAQ contains 14 questions & 3 subscales (Educational, Relational, & Psychological functioning) embedded within. Each subscale is scored on 1(very inaccurate)-5 (very accurate) likert scale. Educational Functioning items include: 1, 5, 7, 12, 13; Relational Functioning items include: 2, 4, 9, 10, 14; Psychological Functioning items include: 3, 6, 8, 11. Items 2 & 9 from Relational subscale, 13 from Educational subscale, & 8 & 11 from Psychological subscale are reversed scored on 5 (very inaccurate)-1(very accurate) likert scale.
  The Educational functioning subscale score can be summed range from 5-25; the Relational functioning subscale score can be summed range from 5-25; the Psychological subscale can be summed range from 4-20. Total scores across all 3 subscales can be summed & range from 14-70. Higher scores indicate better functioning on each scale and across the total measure.
Time Frame: 1 month timepoint
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 32 | 17
score on a scale
  Educational Functioning | 21.0 (4.8) | 19.4 (4.0)
  Psychological Functioning | 14.3 (4.1) | 12.1 (4.0)
  Relational Functioning | 17.7 (5.3) | 14.5 (6.2)

13. Secondary Outcome: Psychosocial Functioning
Description: as for outcome 12
Time Frame: 2 month timepoint
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 32 | 15
score on a scale
  Educational Functioning | 20.2 (4.6) | 17.7 (5.6)
  Psychological Functioning | 14.3 (4.3) | 10.8 (3.9)
  Relational Functioning | 17.3 (5.2) | 13.7 (5.6)

14. Secondary Outcome: Psychosocial Functioning
Description: as for outcome 12
Time Frame: 3 month timepoint
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 31 | 14
score on a scale
  Educational Functioning | 21.0 (4.1) | 18.0 (6.5)
  Psychological Functioning | 14.2 (3.8) | 10.1 (4.1)
  Relational Functioning | 17.1 (5.1) | 13.1 (6.4)

15. Secondary Outcome: Symptom Severity
Description: Symptom severity will be assessed via the CCAPS Mental Health Symptoms. The CCAPS is a 62-item instrument with 8 subscales (depression, general anxiety, social anxiety, academic distress, eating concerns, family distress, hostility, substance abuse) related to psychological symptoms & distress in college students. Scores are on a 5 point likert scale for each subscale: 0 (not at all like me), 1,2,3,4 (Extremely like me). Lower scores indicate greater severity of symptoms. Some items are reverse-scored. To score, average the items scores for each subscale to create the subscale raw score.
Time Frame: 1 month timepoint
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 32 | 17
score on a scale
  Depression | 1.36 (0.96) | 1.57 (1.00)
  General Anxiety | 1.82 (1.05) | 2.02 (1.07)
  Social Anxiety | 2.06 (1.07) | 2.15 (0.95)
  Academic Distress | 1.45 (1.06) | 1.76 (0.96)
  Eating Concerns | 1.22 (1.03) | 1.61 (1.11)
  Family Distress | 1.13 (0.96) | 1.41 (1.00)
  Hostility | 0.93 (0.80) | 1.26 (0.81)
  Substance Abuse | 0.43 (0.72) | 0.32 (0.54)

16. Secondary Outcome: Symptom Severity
Description: as for outcome 15
Time Frame: 2 month timepoint
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 32 | 15
score on a scale
  Depression | 1.24 (0.94) | 1.85 (1.02)
  General Anxiety | 1.70 (1.15) | 2.24 (0.99)
  Social Anxiety | 1.92 (1.07) | 2.39 (1.02)
  Academic Distress | 1.39 (1.06) | 2.13 (0.90)
  Eating Concerns | 1.21 (0.97) | 1.72 (1.13)
  Family Distress | 1.18 (0.82) | 1.13 (0.83)
  Hostility | 0.75 (0.82) | 1.39 (0.86)
  Substance Abuse | 0.38 (0.60) | 0.21 (0.38)

17. Secondary Outcome: Symptom Severity
Description: as for outcome 15
Time Frame: 3 month timepoint
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 31 | 14
score on a scale
  Depression | 1.12 (0.94) | 1.83 (1.11)
  General Anxiety | 1.42 (0.99) | 1.96 (0.93)
  Social Anxiety | 1.81 (1.03) | 2.39 (0.90)
  Academic Distress | 1.31 (0.98) | 2.12 (1.11)
  Eating Concerns | 1.01 (0.86) | 1.55 (0.97)
  Family Distress | 0.93 (0.63) | 1.10 (0.71)
  Hostility | 0.82 (0.89) | 1.10 (0.73)
  Substance Abuse | 0.40 (0.58) | 0.39 (0.76)

18. Secondary Outcome: Mental Health Service Follow-through
Description: Mental health service follow-through will be assessed via the Client Service Receipt Inventory (CSRI). Ratings of 4 questions are Yes or No indicating if participants received the type of service. Scores described below are count of participants indicating "Yes" on the scale.
Time Frame: 1 month timepoint
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 32 | 17
Participants
  Any mental health care | 17 | 11
  Inpatient | 0 | 0
  Outpatient | 15 | 11
  Primary care | 4 | 1

19. Secondary Outcome: Mental Health Service Follow-through
Description: as for outcome 18
Time Frame: 2 month timepoint
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 32 | 15
Participants
  Any mental health care | 16 | 11
  Inpatient | 0 | 1
  Outpatient | 12 | 10
  Primary care | 6 | 3

20. Secondary Outcome: Mental Health Service Follow-through
Description: as for outcome 18
Time Frame: 3 month timepoint
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
Number analyzed (Participants) | 31 | 14
Participants
  Any mental health care | 15 | 7
  Inpatient | 0 | 0
  Outpatient | 12 | 7
  Primary care | 5 | 1

ADVERSE EVENTS:
Time Frame: Participant level information was assessed for adverse events at each of 3 follow up timepoints (1 month, 2 months, and 3 months after baseline).
Arm/Group | Text2Connect Intervention | Usual Care-Psychoeducational Videos (PE) Only
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/18
Other Adverse Events (participants affected / at risk) | 0/34 | 0/18

LIMITATIONS AND CAVEATS:
Findings may not be valid in men or racial or ethnic minorities due to makeup of sample. This study may have a limited understanding of durability, prolonged engagement, and typical experiences and stresses related to college transition due to only following participants for 3 months during COVID pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT04560075/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT04560075/ICF_001.pdf